CLINICAL TRIAL: NCT04076592
Title: Children Nutrition as a Protective or Health-risk Factor
Brief Title: NUTRIPROTECT-Children Nutrition as a Protective or Health-risk Factor
Acronym: My-Milk-2
Status: Completed | Type: Observational
Sponsor: University of Ljubljana (Other)
Collaborators: University Medical Centre Ljubljana (Other)
Responsible Party: Sponsor
Other Study IDs: L3 8213 BF-UL My-Milk-2
Record Dates: First submitted 2019-07-30; First posted 2019-09-03 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-09

CONDITIONS: Breastfeeding; Dietary Intake; Health; Body Composition; Intestinal Microbiota
Keywords: Nutritional Intake,; Child Growth and Development; Bone Density; Antibiotics
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — child's feces
Oversight: Data Monitoring Committee: No

SUMMARY:
Despite the intensive worldwide research dedicated to the nutrition and faecal microbiota, the studies that follow the link between the early nutrition, initial intestinal microbiota, and development of children over a longer time period are limited. From 2010 to 2013, the investigators conducted a study "My-Milk" in Slovenia. From 185 participating pregnant women involved in the detailed part of the protocol (comprising of 4-days weighed dietary record, visits at clinic and biological sample collection), 152 participants completed the study at the child's first year of age. Five of the participants bore twins whose data was excluded from the research because infant's identity was not consistently followed throughout the research. In addition to studying the microbiota and fatty acid composition of breast milk and the initial development of intestinal microbiota of breastfed babies, the investigators also monitored the diet of expecting and nursing participants, concentration of vitamin D in serum and bone mineral density in participating mothers and children. The investigators performed anthropometric measurements of children during the first year of age. All singleton children who have completed My-Milk study (N= 147) will be invited in the follow-up study "My-Milk-2". The first step of the proposed study will be the evaluation of nutritional status of children aged 6 to 7 years in 2017/2018, including the assessment of the body composition (bone density, percentage of fat and muscle tissue), health indicators (blood pressure, blood cholesterol, frequency and severity of infections) and fecal microbiota. The obtained data of My-Milk and My-Milk-2 studies will enable the prospective cohort study to be carried out on the effects of early nutrition and various factors of mother and child during the first year of age on the health and developmental status of children aged 6- 7 years. The project results will significantly improve the progress in research areas of public health and nutrition. The interactions along the axis nutrition in early childhood, gut microbiota composition/ diversity and potential health problems in later life are still not fully explored. The investigators expect the results of the proposed study will contribute to the scientific development in this field in global prospective. The acquired information will also be an excellent basis for development of new dietary guidelines for children.

DETAILED DESCRIPTION:
Nutrition can act either as a risk or protective factor in the development of a series of non-communicable diseases. While such effects were established for the whole life cycle, the nutrition in early life may be particularly relevant for its long-term impact on later life health. The reliable scientific data on dietary intakes and nutritional status of the representing sample population serve as a basis to elucidate the role, the specific nutritional factors exert on human health. The scientific background of the proposed applicative research project is based on the fact that the studies, following the link between the early nutrition, initial intestinal microbiota, and development of children, over a longer time period, are limited. Therefore, the key scientific challenges addressed are focused on the effects of the early life nutrition on growth and health of participating children, and to investigate the relationship among various markers of health.

While the work programme of this multidisciplinary applicative prospective study will be focused onto children, it shall be tightly linked to former "My-Milk" project (SRA J43606; finished in the year 2013), where the role of early nutrition in the development of breast fed children and their intestinal microbiota, during the first year of life, was investigated. This study will be conducted within the population of 6-7 years olds included in the first "My-Milk" study. The study will characterize the key modifying factors during participant's early life (defined through maternal variables (BMI before pregnancy, weight gain during pregnancy, nutrition during pregnancy and lactation, fatty acid composition of human milk, and vitamin D concentration in serum) and infant variables (duration of breastfeeding and antibiotic treatments, faecal microbiota at first month, anthropometrics and bone mineral density in the neonatal period)) on participant's nutritional status at the age 6-7 years. The current nutritional status will be defined by participant's dietary intakes, anthropometrics, body composition - bone density, percentage of fat and muscle tissue), health (blood pressure, blood cholesterol, frequency and severity of infections), and fecal microbiota.

The study population invited to participate will include all singleton children of mothers who completed the detailed part of the My-Milk study at child's first year of age (N=147). Considering a very low drop-out rate in the first detailed part of the study My-Milk (33 participating mothers out of 185, approximately 18 percent), investigators expect that at least 70-75 percentage of the invited participants will respond, meaning between 100 - 110 children may get enrolled in the study. This population will represent 0,5 percentage of children born in 2011 (21947 children - statistical data for Slovenia).

The following parameters will be measured and evaluated: the nutrition of children by using the standard dietary assessment methodology for children and adults/elderly population as provided in the European Food Safety Authority guidance (EFSA). Namely, the food consumption survey will be carried out on the individual level by repeated 24-h food diary and Computer Assisted Personal/Telephone Interview method (CAPI/CATI) and by supporting General Questionnaire and the Food Propensity Questionnaire (FPQ) according to PANCAKE - Pilot study for the Assessment of Nutrient intake and Food Consumption Among Kids in Europe. The 24-h structured diet recall interview is a quantitative research method used in the nutritional assessment. A trained dietitian investigator will ask a parent or caretaker to recall all foods and drinks that the participating child consumed during the previous 24 hours at two different time points during the study (non-consecutive days at least 8 - 20 days between the two records) to receive the proper information about the habitual intake of foods. From the data obtained by 24-h recall investigators intend to evaluate nutritional intakes of the population sub-groups. In addition, connections between the nutrition of children and body composition and health markers will be studied. FPQ will enable the estimation of certain relevant, infrequently consumed food groups. Data will be collected using validated questionnaires using computer -assisted data collection methods and processing. Evaluation of the dietary intake data will be performed by dietary software Open Platform for Clinical Nutrition (OPEN) by Jožef Stefan Institute (IJS). OPEN is a web-based application for dietary assessment and treatment as well as upgraded to support the 24h -recall/food diary method and FPQs in line with the EFSA pan-European food consumption survey, also known as the EU Menu, methodology. OPEN is an efficient, first Slovenian web-based tool for dietary assessment based on the local food items. OPEN allows the dietitian to enter the food and amounts for each participant. After food items, amounts and preparations are entered into the OPEN, the program creates an analysis with the breakdown of nutritional information.

The assessment of growth, development, and health status in 6-7 years old participants will base on the conducted clinical examination and data obtained from the medical records. Clinical examination will include the assessment of clinical status, anthropometric measurements, and quantitative ultrasound measurements of the bone mineral density and measurement of blood pressure.

The clinical examination will be performed at the University Children's Hospital and will be carried out by a specialist doctor of paediatrics and investigator biologist. It will include the assessment of clinical status, anthropometric measurements, and quantitative ultrasound measurements of bone mineral density. The bone mineral density will be measured at the right tibia using the (QUS) Sunlight Omnisense (Sunlight Medical Ltd, Tel Aviv, Israel) which is simple, painless and radiation free investigation and gives information about the bone density and micro architecture. The QUS measures the time taken by the ultrasound signal to travel between two transmitters and two receivers contained within the probe. These propagation times are used by a proprietary algorithm to determine the bone speed of sound (SOS), which is expressed as meters per second (m/s). The software will use the three most consistent measurements to compute the result. The results will be taken as SOS and Z score (units of standard deviations relative to the mean for age- and sex-matched population reference values). Unlike in children, in adults, measurements are taken on a radius. For anthropometry: body height [cm] and body mass [kg] will be measured with a certified medical scale barefooted and in a minimal clothing. The precision of a height measurement will be 0.1 cm and of a mass measurements 0.1 kg. Skinfold thicknesses [mm] at six standard locations will be measured according to the standardised methodology with the precision of 0.1 mm by a calibrated certified skinfold calliper (Harpenden, England). Circumferences [cm] will be measured once on the trunk or on the right side of the body with a non-stretchable narrow measuring tape (fibre glass tape, China) with the precision of 0.1 cm. The estimates of body composition will be linked to the acquired nutritional data.

Other information regarding the current health status (including blood cholesterol) and child development will be obtained from the medical documentation. For this purpose investigators will ask paediatricians for the access to the participants' medical records. The data on the eventual disruption of a regular physical development shall be analysed (the accelerated growth, attenuated growth, low body mass and BMI for overweight or obesity), and on the presence of allergies and emerging chronic diseases. The emphasis will also be laid on the infections, medication intakes (antibiotic treatments) and chronic diseases.

The study of children fecal microbiota will base on molecular approaches such as quantitative real-time PCR (qPCR) and next-generation sequencing (NGS) sequencing of the 16 sedimentation coefficient (16S) subunit of ribosomal ribonucleic acid (rRNA) gene amplicons using Illumina technology. A single fecal sample of an apparently healthy child will be collected at the clinical examination. Priorly, the parents will be supplied with the coded sterile sampling containers with a spoon attached to the lid and with sampling instruction by post and e-mail. They will be asked to collect approximately 2 g (2 spoons) of participating child's faeces possibly on the planned day of visit at the Pediatric clinic or one day before. Samples will be kept refrigerated/cooled until the visit and will be immediately frozen at -20 ˚C upon the arrival to the clinic by the medical personnel. Within a month after being collected, -20 ˚C frozen fecal samples will be transferred to the laboratory and stored at -80 ˚C until the performance of microbial analyses. QPCR and 16S rRNA amplicon sequencing methods, also applied in the first part of My-Milk project, are suitable for the assessment of the biodiversity among total bacterial communities and composition of fecal microbiota, as well as, the evaluation of the quantitative fluctuations of specific target groups in the complex microbial ecosystems such as gastrointestinal tract.

Data about the nutrition of 6-7-year old participants will be studied in connection with body composition (bone density, fat percentage, and muscle tissue), health markers (blood pressure, blood cholesterol), and fecal microbiota. After quality control of the sequenced reads, the faecal microbiome biodiversity and relative abundance of bacterial taxa will be gained and biodiversity measures such as the Chao1 score and the Shannon diversity index will be calculated.

Afterwards, all data will be deposited in the central database together with those already obtained during the first part of My-Milk study. The appropriate statistical analysis will be applied in investigating the impact of early life exposures on later growth, nutritional status, health and faecal microbiota in participants at the current age of 6-7 years. The central database will allow (a) protected access to already collected information; (b) addition of new attributes and (c) export of data for the purposes of statistical analysis. Database will not contain any personal identifications (subjects will be coded by identification numbers only). The majority of the collected data from My-Milk study have already been converted into electronic form. Statistical methodology will comprise of the two steps: the first exploratory step, which consists of the data checking, graphical displays and reduction of higher dimensional space into lower dimensional space via multivariate statistical methods, such as principal component analysis and multivariate scaling; the second step will be devoted to statistical inference. The appropriate statistical tests will be used, regression models will be derived taking into account the research hypotheses. The power of the tests will be calculated and the models will be critically assessed by modern simulation techniques (e. g. bootstrap approach).

ELIGIBILITY:
Inclusion Criteria:

* all singleton children and their mothers who have completed a detailed part of the My-Milk study (N=147) will be invited in this follow-up study.

Exclusion Criteria: /

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: All singleton children and their mothers who have completed a detailed part of the My-Milk study 1 (147) will be invited in this prospective follow-up study.
Sampling Method: Non-Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-01-11 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
Assessment of Nutritional Status of Children Using Dietary Pattern- Energy Intake | through study completion, an average of 1 year
  Habitual energy intake per day in kilocalories (kcal): calculated online with the software OPEN platform having integrated Slovenian food database, from child's 24-hour dietary recalls (of food items ingested) on two non-consecutive days.
Assessment of Nutritional Status of Children Using Dietary Pattern- Average Nutrient Intake | through study completion, an average of 1 year
  An average intake of carbohydrates, total sugar, free sugar, starch, dietary fibres, fat, fatty acids, proteins per day in percentages: calculated online with the software OPEN platform having integrated Slovenian food database, from child's 24-hour dietary recalls (of food items ingested) on two non-consecutive days.
Assessment of Nutritional Status of Children Using Dietary Pattern- Average Intake of eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA) | through study completion, an average of 1 year
  An average intake of adjusted eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA) per day in grams: calculated online with the software OPEN platform having integrated Slovenian food database, from child's 24-hour dietary recalls (of food items ingested) on two non-consecutive days.
Assessment of Nutritional Status of Children Using Dietary Pattern- Adjusted Intake of Vitamin D | through study completion, an average of 1 year
  An adjusted vitamin D and folic acid intake per day in micrograms: calculated online with the software OPEN platform having integrated Slovenian food database, from child's 24-hour dietary recalls (of food items ingested) on two non-consecutive days.
Assessment of Nutritional Status of Children Using Dietary Pattern- Adjusted Micronutrients Intake | through study completion, an average of 1 year
  An adjusted natrium, chlorine, calcium and iron in milligrams: calculated online with the software OPEN platform having integrated Slovenian food database, from child's 24-hour dietary recalls (of food items ingested) on two non-consecutive days.
Assessment of Nutritional Status of Children Using BMI | through study completion, an average of 1 year
  Body Mass Index calculated from weight/height^2 in kg/m^2.
Assessment of Nutritional Status of Children Using Anthropometric Measurements - Sitting Height, Leg Length and Circumferences | through study completion, an average of 1 year
  Sitting height, leg length -iliospinal, circumference for upper arm, waist, calf in cm.
Assessment of Nutritional Status of Children Using Anthropometric Measurements- Skinfold Thickness | through study completion, an average of 1 year
  Skinfold thickness for biceps, triceps, subscapular, iliac crest, calf in mm.
Assessment of Nutritional Status of Children Using Bone Density Measurements | through study completion, an average of 1 year
  Bone density in meters per second expressed as units of standard deviations relative to the mean for age- and sex-matched population reference values.
Nutritional Status of Children Using Systolic and Diastolic Blood Pressure | through study completion, an average of 1 year
  Systolic and Diastolic Blood pressure in mmHg;
Assessment of Nutritional Status of Children Using Blood Cholesterol | through study completion, an average of 1 year
  Blood cholesterol in mg/dL
Assessment of Nutritional Status of Children Using Morbidity (Sickness Frequency) | through study completion, an average of 1 year
  Frequency of infections and consumed antibiotics.
Assessment of Nutritional Status of Children Using Fecal Microbiota | through study completion, an average of 1 year
  Fecal microbiota composition (expressed in percentages of relative abundances of represented amplicons of bacterial groups).

SECONDARY OUTCOMES:
Changes in BMI from first year till 7th year of life | from first year data till 7th year of life
  Changes in BMI-weight/height^2 in kg/m^2 (expressed as units of standard deviations relative to the mean for age- and sex-matched population reference values)
Changes in Bone Density from first year till 7th year of life | from first year data till 7th year of life
  Changes in bone density in meters per second (expressed as units of standard deviations relative to the mean for age- and sex-matched population reference values).
Correlation Early Feeding and BMI at age 7 years | through study completion, an average of 1 year
  Correlations (expressed as Spearman, Pearson, etc. coefficients) in association study between the type of early feeding (exclusive breastfeeding vs formula supplementation) and BMI-weight/height^2 in kg/m^2.
Correlation Between Breastfeeding Length and BMI at age 7 years | through study completion, an average of 1 year
  Correlations (expressed as Spearman, Pearson, etc. coefficients) in association study between the length of breastfeeding (in months) and BMI- weight/height^2 in kg/m^2.
Correlation Between Breastfeeding Length and Bone Density at age 7 years | through study completion, an average of 1 year
  Correlations (expressed as Spearman, Pearson, etc. coefficients) in association study between the length of breastfeeding (in months) and bone density in meters per second.
Correlation Between Frequency of Infections and Fecal Microbiota at age 7 years | through study completion, an average of 1 year
  Correlations (expressed as Spearman, Pearson, etc. coefficients) in association study between frequency of infections and fecal microbiota composition.

CONTACTS AND LOCATIONS:
Overall Officials: Irena Rogelj, Prof., PhD, Principal Investigator — University of Ljubljana; Rok Orel, MD, Prof., PhD, Study Director — University Medical Centre Ljubljana, Division of Pediatrics
Locations (1):
- University Medical Centre Ljubljana, Division of Paediatrics, Department of Neonatology, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Undecided
Scientific articles

REFERENCES:
- [Background] Dodd KW, Guenther PM, Freedman LS, Subar AF, Kipnis V, Midthune D, Tooze JA, Krebs-Smith SM. Statistical methods for estimating usual intake of nutrients and foods: a review of the theory. J Am Diet Assoc. 2006 Oct;106(10):1640-50. doi: 10.1016/j.jada.2006.07.011. PMID 17000197
- [Background] Subar AF, Dodd KW, Guenther PM, Kipnis V, Midthune D, McDowell M, Tooze JA, Freedman LS, Krebs-Smith SM. The food propensity questionnaire: concept, development, and validation for use as a covariate in a model to estimate usual food intake. J Am Diet Assoc. 2006 Oct;106(10):1556-63. doi: 10.1016/j.jada.2006.07.002. PMID 17000188
- [Background] Farmer G. Neonatal skinfold thickness. Measurement and interpretation at or near term. Arch Dis Child. 1985 Sep;60(9):840-2. doi: 10.1136/adc.60.9.840. PMID 4051541
- [Result] Obermajer T, Grabnar I, Benedik E, Tusar T, Robic Pikel T, Fidler Mis N, Bogovic Matijasic B, Rogelj I. Microbes in Infant Gut Development: Placing Abundance Within Environmental, Clinical and Growth Parameters. Sci Rep. 2017 Sep 11;7(1):11230. doi: 10.1038/s41598-017-10244-x. PMID 28894126
- See also: OPEN: Open Platform for Clinical Nutrition, Available 04.03.2015 — http://www.opkp.si/en_GB/cms/vstopna-stran
- See also: Zekan et al. (1999): Predictive factors in determination of newborn weight — https://hrcak.srce.hr/20334